CLINICAL TRIAL: NCT05228366
Title: The Effect of Heel Warming With Mild and Hot Thermofor Applied Before Heel Lance on Total Crying Time and Procedure Time in Healthy Term Newborns.: A Randomized Clinical Trial
Brief Title: Heel Warming With Mild and Hot Thermofor Applied Before Heel Lance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isparta University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IspartaUASNursingCare2
Record Dates: First submitted 2022-01-12; First posted 2022-02-08 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2022-02

CONDITIONS: Nursing Caries
Keywords: Heel warming; Heel Lance; Newborn; Total crying time; Processing time

STUDY DESIGN:
Intervention Model Description: 3-armed randomized controlled trial
Who Masked: Participant
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heel warming with mild thermofor group (Experimental): Heel warming will be applied to the newborns in the ıntervention group 1 with a thermofor containing 34-37C warm water for 5 minutes before the heel blood collection procedure. During the procedure, the general condition of the newborn and the changes in his skin will be observed closely. Heel blood collection will be performed by following the standard procedure steps that are routinely applied in the service.
  Interventions: Other: Heel warming with mild thermofor group
- Heel warming with hot thermofor group (Experimental): Heel warming will be applied to the newborns in the ıntervention group 2 with a thermofor containing 38-40C warm water for 5 minutes before the heel blood collection procedure. During the procedure, the general condition of the newborn and the changes in his skin will be observed closely. Heel blood collection will be performed by following the standard procedure steps that are routinely applied in the service.
  Interventions: Other: Heel warming with hot thermofor group
- Ineffective heel warming with thermofor group (Other): Ineffective heel warming will be applied to the newborns in the control group with a thermofor containing 28C warm water for 5 minutes before the heel blood collection procedure. During the procedure, the general condition of the newborn and the changes in his skin will be observed closely. Heel blood collection will be performed by following the standard procedure steps that are routinely applied in the service.
  Interventions: Other: Ineffective heel warming with thermofor group

INTERVENTIONS:
Other: Heel warming with mild thermofor group — Heel warming will be applied to the newborns in the ıntervention group 1 with a thermofor containing 34-37C warm water for 5 minutes before the heel blood collection procedure. During the procedure, the general condition of the newborn and the changes in his skin will be observed closely. Heel blood collection will be performed by following the standard procedure steps that are routinely applied in the service
  Arms: Heel warming with mild thermofor group
Other: Heel warming with hot thermofor group — Heel warming will be applied to the newborns in the ıntervention group 2 with a thermofor containing 38-40C warm water for 5 minutes before the heel blood collection procedure. During the procedure, the general condition of the newborn and the changes in his skin will be observed closely. Heel blood collection will be performed by following the standard procedure steps that are routinely applied in the service
  Arms: Heel warming with hot thermofor group
Other: Ineffective heel warming with thermofor group — Ineffective heel warming will be applied to the newborns in the control group with a thermofor containing 28C warm water for 5 minutes before the heel blood collection procedure. During the procedure, the general condition of the newborn and the changes in his skin will be observed closely. Heel blood collection will be performed by following the standard procedure steps that are routinely applied in the service.
  Arms: Ineffective heel warming with thermofor group

SUMMARY:
Heel warming with thermophor during heel blood collection is a cost-effective and easy-to-apply method. In previous studies, it has been shown that applying heat to the heel reduces the pain of taking heel blood, increases comfort and shortens the procedure time and total crying time. Warm aplication increases the skin surface temperature, causing proximal vasodilation, thereby accelerating blood flow and increasing blood circulation. Increased blood circulation can reduce the pressure applied to the heel of newborns, shorten the procedure time, reduce the perception of pain and increase comfort. As a result of the literature review, it is seen that there is no clarity about the temperature degrees used in heel heating. It has been seen in the literature that warming the heel before heel blood collection is often carried out as mild (34-37C) or hot (38-40C). This study aims to determine heel warming with mild (34-37C) and hot (38-40C) thermofor applied before heel lance on total crying time and procedure time in healthy term newborns.

DETAILED DESCRIPTION:
Aim: The effect of heel warming with mild (34-37C) and hot (38-40C) thermofor applied before capillary heel blood sampling on total crying time and procedure time in term newborns.

Method: This study was planned as a randomized controlled, experimental, double-blind, single-center study. The universe of the research will be term newborns whose heel blood samples will be taken within the scope of the Newborn Screening Program (NSP) in the Isparta Şehir Hospital Gynecology and Obstetrics III Service.

The sample of the study was determined as 120 healthy term newborn (40 control, 40 intervention 1, 40 intervention 2).

Intervention: In this study, ineffective heel warming with thermofor will be applied to the control group; heel warming with mild (34-37C) thermofor will be applied to the intervention group 1; heel warming with hot (38-40C) thermofor will be applied to the intervention group 2. All newborns will breastfed from their mothers during and after the procedure.

Data collection instruments: Newborn Information Form (NIF).

Data collection: Heel blood collection will be video-recorded from the pre-evaluation stage (one minute before the intervention) until the 5th minute after the puncture heel. The video recording will be monitored by independent evaluator who do not know the purpose of the study, and the processing time will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Born between 38-42 gestational weeks (term newborns)
* Newborns with a birth weight of 2500-4400 grams
* Newborns with stable physiological parameters and general condition
* Newborns with vitamin K and hepatitis B vaccine in the delivery room
* Newborns with eight or more Apgar scores in the first and fifth minutes

Exclusion Criteria:

* Newborns with problems during pregnancy, labor and postpartum
* Newborns with congenital anomaly
* Newborns receiving pharmacological or non-pharmacological pain management intervention before the procedure
* Newborns with receiving oxygen therapy
* Newborns with having undergone a surgical procedure
* Newborns with sepsis or suspected sepsis
* Newborns whose parents state that they want to leave the study while the study continues

Ages: 24 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Prosedüre time measure | During the procedure
  The video recording will be monitored by independent evaluator who do not know the purpose of the study, and the processing time will be recorded.

SECONDARY OUTCOMES:
Total crying time | Up to 5 minutes after the heel stick
  The video recording will be monitored by independent evaluator who do not know the purpose of the study, and the total crying time will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Fahriye PAZARCIKCI, Study Director — Isparta University of Applied Sciences, Isparta, Turkey
Locations (1):
- Isparta University of Applied Sciences, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
N/O

REFERENCES:
- [Background] Shu SH, Lee YL, Hayter M, Wang RH. Efficacy of swaddling and heel warming on pain response to heel stick in neonates: a randomised control trial. J Clin Nurs. 2014 Nov;23(21-22):3107-14. doi: 10.1111/jocn.12549. Epub 2014 Jan 30. PMID 24476226